CLINICAL TRIAL: NCT00126880
Title: A Phase II, Randomised, Double-blind, Dose-ranging Study of AVX754 Versus Lamivudine in Treatment-experienced HIV-1 Infected Patients With the M184V Mutation in Reverse Transcriptase
Brief Title: AVX754 (a New Nucleoside Reverse Transcriptase Inhibitor [NRTI]) to Treat Drug-resistant HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avexa (Industry)
Responsible Party: Susan Cox, Avexa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVX-201
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus; anti-retroviral therapy; nucleoside analogue; reverse transcriptase; lamivudine; resistance mutation; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — apricitabine; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 600mg BID ATC (Experimental): 600mg BID ATC
  Interventions: Drug: AVX754
- 800mg BID ATC (Experimental): 800mg BID ATC
  Interventions: Drug: AVX754
- 150mg BID 3TC (Active Comparator): 150mg BID 3TC
  Interventions: Drug: 3TC

INTERVENTIONS:
Drug: AVX754 — apricitabine, 600mg BID or 800mg BID
  Other Names: apricitabine
  Arms: 600mg BID ATC; 800mg BID ATC
Drug: 3TC — 3TC, 150mg BID
  Other Names: lamivudine
  Arms: 150mg BID 3TC

SUMMARY:
The study will measure how safe and effective AVX754 (a new drug for the treatment of HIV) is in treating HIV-1 infected people who have failed treatment with lamivudine.

DETAILED DESCRIPTION:
Lamivudine or emtricitabine are commonly used in combination with other drugs for first-line treatment of HIV infection. Although effective initially, many people later on develop resistance to some or all of the drugs (including lamivudine) leading to virological failure. Resistance is associated with characteristic mutations, which for lamivudine is the M184V mutation. A change to new, active drugs must take place when patients fail their current regime, to regain control of the virus. Although there are other types of drugs available for second line treatment, there is currently no fully active, well tolerated cytidine analogue that can replace lamivudine in a second-line regimen when patients fail first line treatment. This study will measure the efficacy and safety of AVX754 (a novel cytidine analogue with activity against HIV resistant to other nucleosides) as part of a new regimen to treat patients who have failed treatment containing lamivudine, compared to the best alternative new regimen which continues to include lamivudine.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* M184V mutation in reverse transcriptase
* Currently taking lamivudine
* Viral load >2000 copies/ml

Exclusion Criteria:

* Hepatitis B surface antigen positive
* Pregnant or breastfeeding females
* Hepatitis C RNA positive and requiring treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV RNA levels at day 21 | day 21
Time-weighted average change from baseline in HIV RNA levels through 21 days | 21 days

SECONDARY OUTCOMES:
Change from baseline in HIV RNA levels at days 7, 14, 21 | days 7, 14, 21
Proportion of subjects with HIV RNA levels <400 or <50 at days 7, 14, 21, and weeks 24 and 48 | days 7, 14, 21, and weeks 24 and 48
Change from baseline and change in ratio of CD4+ and CD8+ cells at day 21 and weeks 24 and 48 | day 21 and weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Cox, Ph D, Study Director — Avexa
Locations (1):
- Avexa (co-ordinating sites in Australia and Argentina), Melbourne, Victoria, Australia